CLINICAL TRIAL: NCT06215196
Title: Effectiveness and Safety of Semaglutide Combined With Dietary Fiber (Soloways) in Adults With Overweight or Obesity: A Randomized, Placebo-Controlled, Double-Blind Clinical Trial
Brief Title: Effectiveness and Safety of Semaglutide Combined With Dietary Fiber (Soloways) in Adults With Overweight or Obesity
Acronym: ESSENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other); Triangel Scientific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW004
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Overweight and Obesity
Keywords: Semaglutide; Weight Loss; Obesity; Appetite Suppression
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide with Active Fiber Supplement Group (Experimental)
  Interventions: Dietary Supplement: Fiber Supplement Group
- Placebo group (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Fiber Supplement Group — Semaglutide (2.4 mg weekly). Three daily packets of active fiber supplement (each containing 1g of glucomannan, 1g of inulin, and 3g of psyllium), taken 30 minutes before each main meal. The supplement is provided by S.Lab (Soloways), LLC.
  Arms: Semaglutide with Active Fiber Supplement Group
Other: placebo — Semaglutide (2.4 mg weekly). Three daily packets of placebo powder, taken 30 minutes before each main meal.
  Arms: Placebo group

SUMMARY:
This clinical trial investigated the combined effects of Semaglutide and a fiber supplement (glucomannan, inulin, psyllium) on weight loss in adults with overweight or obesity. Participants, aged 18-65 with a BMI ≥30 or ≥27 with comorbidities, were randomized into two groups: one receiving Semaglutide with active fiber supplements and the other with Semaglutide and placebo, over a 180-day period. Key endpoints included percentage change in body weight, BMI, body composition, safety, and appetite control, with a focus on evaluating the additive effects of dietary fibers in enhancing Semaglutide's efficacy.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30, or ≥27 with comorbidities.

Exclusion Criteria:

* Serious chronic illnesses.
* History of bulimia or anorexia.
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline | 180 days
Achievement of a reduction in body weight of 5% or more from baseline. | 180 days

SECONDARY OUTCOMES:
BMI change | 180 days
fat mass change | 180 day
  fat mass change assessed using bioelectrical impedance analysis
Safety evaluated by recording any adverse events. | 180 days
fat-free mass change | 180 days
  fat-free mass change assessed using bioelectrical impedance analysis
visceral fat rating change | 180 days
  visceral fat rating change assessed using bioelectrical impedance analysis
total body water change | 180 days
  total body water change assessed using bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia